CLINICAL TRIAL: NCT03521778
Title: Fascial Distortion Model Manual Therapy and Painful Shoulder Syndrome
Acronym: FDM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Józef Piłsudski University of Physical Education (Other)
Responsible Party: Principal Investigator, Adrian Rogala, PhD Student, Józef Piłsudski University of Physical Education
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JozefPilsudskiU
Record Dates: First submitted 2018-04-15; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-04

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fascial Distortion Model group (Experimental): Patients will receive manual treatment complies with Fascial Distortion Model method.
  Interventions: Other: Fascial Distortion Model
- Mulligan Concept group (Experimental): Patients will receive manual treatment complies with Mulligan Concept method.
  Interventions: Other: Mulligan Concept
- Traditional physiotherapy group (Experimental): Patients will receive traditional physiotherapy.
  Interventions: Other: Traditional physiotherapy

INTERVENTIONS:
Other: Fascial Distortion Model — Patients will receive manual treatment according to FDM procedures:
  1. Triggerbands - therapist put a pressure by the thumb along the presented pathway.
  2. Continuum Distortions - therapist put a pressure by the thumb at the exact place of feeling of pain.
  3. Folding Distortions - therapist conduct traction or compression of the affected joint.
  4. Herniated Triggerpoint - therapist put a pressure by the thumb at the place where HTP occurs.
  5. Cylinder Distortions - therapist compress and stretch by the hands affected area.
  6. Tectonic Fixation - Therapist compress and stretch affected area by the hands or tools like vacuum bubble.
  Other Names: Manual treatment- Fascial Distortion Model
  Arms: Fascial Distortion Model group
Other: Mulligan Concept — Patients will receive manual treatment according to Mulligan Concept procedures:
  MWM- Mobilization With Movement- application can be defined as the application of a sustained passive force/glide.
  NAG - Natural Apophyseal Glide - application can be defined as the oscillatory mobilization techniques from the middle to the end of the range of motion.
  SNAG- Sustained Natural Apophyseal Glide- They are weight bearing techniques: all procedures are done with the patient sitting or in standing. They are mobilisations with active movement followed by passive over pressure.
  Other Names: Manual treatment- Mulligan Concept
  Arms: Mulligan Concept group
Other: Traditional physiotherapy — Patients will receive traditional physiotherapy:
  Exercises, laser treatment, magnetic field therapy, ultrasound treatment, light treatment
  Arms: Traditional physiotherapy group

SUMMARY:
Relatively new method of diagnosing and treating dysfunction of the musculoskeletal system is Fascial Distortion Model. It is manual therapy developed by emergency physician and an osteopath Stephen P. Typaldos.

Disfunction are diagnosed based on verbal and physical descriptions, palpations, anamnesis. As a result of examination, It can be found one or more of six different distortions. The aim of the study is to examine the effectiveness of FDM manual therapy in comparison to manual therapy using the Mulligan Concept method and traditional physiotherapy in patients with shoulder dysfunction who have undergone previous rehabilitation and who have not achieved satisfactory results. Patients will receive five treatments with one day brake between each treatment. The patient's condition will be evaluated before the first treatment, two weeks after the last treatment, and also after three months. As a outcome of the occurring phenomenon, structural changes are planned at the level of the fascial system in the studied region. The obtained results may influence the current views on diseases of the musculoskeletal system, as well as on the method of diagnosing and treating shoulder joint dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of dysfunction in the shoulder joint based on an orthopedic and/or physiotherapeutic examination confirmed by X-ray and ultrasound imaging,
* patients undergoing prior rehabilitation / pharmacotherapy / surgical intervention without satisfactory results,
* limitation of mobility and / or pain in the shoulder complex,

Exclusion Criteria:

* coexistence of neoplastic diseases,
* symptoms from the cervical spine
* pregnancy,
* aneurysms,
* osteitis,
* arthritis
* deep veins thrombosis of upper limbs,
* resignation from the study / therapy,
* skin damage, hematomas.

Ages: 40 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-05-25 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline DASH Outcome Measure at 3 months | 1'st day, 2 weeks after treatment, 3 months after treatment
  The Disabilities of the Arm, Shoulder and Hand (DASH) Outcome Measure is a 30-item, self-report questionnaire designed to measure physical function and symptoms in patients with any or several musculoskeletal disorders of the upper limb. It helps describe the disability experienced by people with upper-limb disorders and also to monitor changes in symptoms and function over time .The DASH is scored in 30 items from 1 to 5. Higher score means greater level of disability.
Change from baseline Constant-Murley Shoulder Outcome Score at 3 months | 1'st day, 3 months after treatment
  The Constant-Murley score (CMS) is a 100-points scale composed of a number of individual parameters. These parameters define the level of pain and the ability to carry out the normal daily activities of the patient.[1] The Constant-Murley score was introduced to determine the functionality after the treatment of a shoulder injury. The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher score, the higher the quality of the function.
Change from baseline Quality Of Life Questionnaire SF- 36v2 at 3 months | 1'st day, 3 months after treatment
  The SF-36 is a 36 item questionnaire that measures eight multi-item dimensions of health: physical functioning (10 items) social functioning (2 items) role limitations due to physical problems (4 items), role limitations due to emotional problems (3 items), mental health (5 items), energy/vitality (4 items), pain (2 items), and general health perception (5 items).
Change from baseline Visual Analogue Scale at 3 months | 1'st day, 3 months after treatment
  Visual analogue scales (score 0-10) are psychometric measuring instruments designed to document the characteristics of disease-related symptom severity in individual patients and use this to achieve a rapid classification of symptom severity and disease control.
  The higher score, indicate greater level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Bartosz Molik, Professor, Study Chair — Józef Piłsudski University of Physical Education

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tesarz J, Hoheisel U, Wiedenhofer B, Mense S. Sensory innervation of the thoracolumbar fascia in rats and humans. Neuroscience. 2011 Oct 27;194:302-8. doi: 10.1016/j.neuroscience.2011.07.066. Epub 2011 Aug 2. PMID 21839150
- [Background] Liljencrantz J, Olausson H. Tactile C fibers and their contributions to pleasant sensations and to tactile allodynia. Front Behav Neurosci. 2014 Mar 6;8:37. doi: 10.3389/fnbeh.2014.00037. eCollection 2014. PMID 24639633
- [Background] Olausson H, Wessberg J, Morrison I, McGlone F, Vallbo A. The neurophysiology of unmyelinated tactile afferents. Neurosci Biobehav Rev. 2010 Feb;34(2):185-91. doi: 10.1016/j.neubiorev.2008.09.011. Epub 2008 Oct 8. PMID 18952123
- [Background] Stecco C, Macchi V, Porzionato A, Duparc F, De Caro R. The fascia: the forgotten structure. Ital J Anat Embryol. 2011;116(3):127-38. PMID 22852442
- [Background] Stecco A, Gesi M, Stecco C, Stern R. Fascial components of the myofascial pain syndrome. Curr Pain Headache Rep. 2013 Aug;17(8):352. doi: 10.1007/s11916-013-0352-9. PMID 23801005
- [Background] Jacobson JA. Shoulder US: anatomy, technique, and scanning pitfalls. Radiology. 2011 Jul;260(1):6-16. doi: 10.1148/radiol.11101082. PMID 21697306
- [Background] Adstrum S, Hedley G, Schleip R, Stecco C, Yucesoy CA. Defining the fascial system. J Bodyw Mov Ther. 2017 Jan;21(1):173-177. doi: 10.1016/j.jbmt.2016.11.003. Epub 2016 Nov 16. PMID 28167173
- [Background] RALSTON HJ 3rd, MILLER MR, KASAHARA M. Nerve endings in human fasciae, tendons, ligaments, periosteum, and joint synovial membrane. Anat Rec. 1960 Feb;136:137-47. doi: 10.1002/ar.1091360208. No abstract available. PMID 14435991
- [Background] Benjamin M. The fascia of the limbs and back--a review. J Anat. 2009 Jan;214(1):1-18. doi: 10.1111/j.1469-7580.2008.01011.x. PMID 19166469
- [Background] Dawidowicz J, Szotek S, Matysiak N, Mielanczyk L, Maksymowicz K. Electron microscopy of human fascia lata: focus on telocytes. J Cell Mol Med. 2015 Oct;19(10):2500-6. doi: 10.1111/jcmm.12665. Epub 2015 Aug 27. PMID 26311620
- [Background] Gillies AR, Lieber RL. Structure and function of the skeletal muscle extracellular matrix. Muscle Nerve. 2011 Sep;44(3):318-31. doi: 10.1002/mus.22094. PMID 21949456
- [Background] Ingber DE, Wang N, Stamenovic D. Tensegrity, cellular biophysics, and the mechanics of living systems. Rep Prog Phys. 2014 Apr;77(4):046603. doi: 10.1088/0034-4885/77/4/046603. PMID 24695087
- [Background] Ingber DE. Tensegrity I. Cell structure and hierarchical systems biology. J Cell Sci. 2003 Apr 1;116(Pt 7):1157-73. doi: 10.1242/jcs.00359. PMID 12615960
- [Background] Najrana T, Sanchez-Esteban J. Mechanotransduction as an Adaptation to Gravity. Front Pediatr. 2016 Dec 26;4:140. doi: 10.3389/fped.2016.00140. eCollection 2016. PMID 28083527
- [Background] Giamberardino MA, Affaitati G, Fabrizio A, Costantini R. Myofascial pain syndromes and their evaluation. Best Pract Res Clin Rheumatol. 2011 Apr;25(2):185-98. doi: 10.1016/j.berh.2011.01.002. PMID 22094195
- [Background] Yung E, Asavasopon S, Godges JJ. Screening for head, neck, and shoulder pathology in patients with upper extremity signs and symptoms. J Hand Ther. 2010 Apr-Jun;23(2):173-85; quiz 186. doi: 10.1016/j.jht.2009.11.004. Epub 2010 Feb 11. PMID 20149960
- [Background] Hudak PL, Amadio PC, Bombardier C. Development of an upper extremity outcome measure: the DASH (disabilities of the arm, shoulder and hand) [corrected]. The Upper Extremity Collaborative Group (UECG). Am J Ind Med. 1996 Jun;29(6):602-8. doi: 10.1002/(SICI)1097-0274(199606)29:63.0.CO;2-L. PMID 8773720
- [Background] Beaton DE, Katz JN, Fossel AH, Wright JG, Tarasuk V, Bombardier C. Measuring the whole or the parts? Validity, reliability, and responsiveness of the Disabilities of the Arm, Shoulder and Hand outcome measure in different regions of the upper extremity. J Hand Ther. 2001 Apr-Jun;14(2):128-46. PMID 11382253
- [Background] Constant CR, Murley AH. A clinical method of functional assessment of the shoulder. Clin Orthop Relat Res. 1987 Jan;(214):160-4. PMID 3791738
- See also: Fascia: The Tensional Network of the Human Body — https://www.kobo.com/us/en/ebook/fascia-the-tensional-network-of-the-human-body
- See also: Fascia, somatics, proprioception and improvement of motion precision — http://ptis.pl/wp/wp-content/uploads/2016/04/Praktyczna-SchleipKurkowski-Powiez-SomatykaPropriocepcja.pdf
- See also: Complexity of the Tensegrity Structure for Dynamic Energy and Force Distribution of Cytoskeleton during Cell Spreading — http://journals.plos.org/plosone/article?id=10.1371/journal.pone.0014392
- See also: Fascial plasticity - a new neurobiological explanation — https://pdfs.semanticscholar.org/4fa0/f27447715ca65e5237eea7d9473dfd14945d.pdf
- See also: Methodology for assessing the quality of life — http://www.ptfarm.pl/pub/File/Farmacja%20Polska/2009/08-2009/10%20%20QOL.pdf